CLINICAL TRIAL: NCT00289874
Title: A Multicenter, Double-Blind, Placebo Controlled, Randomized, Parallel-Group Study to Evaluate the Clinical Effect of Oral Montelukast Versus Placebo in Persistent Asthma Which is Also Active During Allergy Seasons in Pediatric Patients With Seasonal Aeroallergen Sensitivity
Brief Title: Montelukast in Pediatric Allergic Asthma (0476-336)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-336; 2006_001
Record Dates: First submitted 2006-02-07; First posted 2006-02-10 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast sodium
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — montelukast 5 mg chewable tablet once daily. Up to 3 weeks of treatment.
  Other Names: MK0476
  Arms: 1
Drug: Comparator: Placebo — Placebo. Up to 3 weeks of treatment
  Arms: 2

SUMMARY:
This is a 3-week study to evaluate FEV1 following treatment with drugs in persistent asthma which is also active during allergy seasons in pediatric patients with seasonal aeroallergen sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, ages 6 to 14 years, with persistent asthma that is also active during allergy season
* Patients must demonstrate positive skin prick tests to seasonally relevant geographic aeroallergens

Exclusion Criteria:

* Patient cannot have any other acute or chronic pulmonary disorder

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Papadopoulos NG, Philip G, Giezek H, Watkins M, Smugar SS, Polos PG. The efficacy of montelukast during the allergy season in pediatric patients with persistent asthma and seasonal aeroallergen sensitivity. J Asthma. 2009 May;46(4):413-20. doi: 10.1080/02770900902847727. PMID 19484680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred three sites in US;
  Prime Therapy: March 2006 to July 2007
Pre-assignment Details: Patients who had unresolved symptoms and signs of an upper respiratory tract infection between Visits 1 and 2, or had evidence of active, clinically significant sinus infection within 1 week of Visit 1 or between Visits 1 and 2, or failed to meet minimum requirement for daytime asthma symptoms and daily β-agonist use were excluded.
Groups:
- Montelukast 5 mg: Montelukast 5 mg chewable tablet orally once daily at bedtime for 3 weeks.
- Placebo: Montelukast matching-image placebo tablet orally once daily at bedtime for 3 weeks.
Period: Overall Study
Arm/Group | Montelukast 5 mg | Placebo
Started | 203 | 218
Completed | 197 | 210
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Did not meet eligibility | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 5 mg | Placebo | Total
Number analyzed (Participants) | 203 | 218 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (2.4) | 10.7 (2.4) | 10.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 90 | 171
  Male | 122 | 128 | 250
Daily β-agonist use [Mean (Standard Deviation); unit: Puffs/Day] | 3.01 (1.77) | 2.72 (1.68) | 2.86 (1.73)
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Liters] | 1.81 (0.57) | 1.84 (0.60) | 1.83 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 3
Description: Percent change from baseline in FEV1, a measure of airway function, at Week 3
Time Frame: Baseline and week 3
Population: The full analysis set population (i.e., includes all patients who had baseline and on-treatment measurements).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Montelukast 5 mg | Placebo
Number analyzed (Participants) | 199 | 208
Percent Change | 9.53 [7.05 to 12.01] | 9.15 [6.71 to 11.59]

2. Secondary Outcome: Percent Change From Baseline in Mean Daily "as Needed" β-agonist Use Over the 3-week Treatment Period
Description: Percent change from baseline in average daily β-agonist use over the 3-week treatment period
Time Frame: Baseline and Week 3
Population: The full analysis set population (i.e., includes all patients who had baseline and on-treatment measurements).
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | Montelukast 5 mg | Placebo
Number analyzed (Participants) | 198 | 212
Percent Change | -18.88 (84.75) | -12.40 (53.88)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during the 6 week, double-blind treatment period, and up to and including 14 days after the last dose of study therapy
Description: The number of participants listed in the SAE table (203 montelukast & 217 placebo) is the number that received treatment.
  Although a participant may have 2 or more AEs they are counted only once in a category. The same participant may appear in other categories.
Arm/Group | Montelukast 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/203 | 4/217
Other Adverse Events (participants affected / at risk) | 0/203 | 0/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 5 mg (N=203) | Placebo (N=217)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Safety is reported in the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.